CLINICAL TRIAL: NCT03829072
Title: Impact of Cooking Education and Adapted Physical Activity on Nutritional Status and Quality of Life of Patients Treated by Allo Stem Cell Transplantation
Brief Title: Cooking Education and Adapted Physical Activity in Allografted Patients
Acronym: NUTRITION
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 18-PP-10
Record Dates: First submitted 2018-12-27; First posted 2019-02-04 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Allograft
Keywords: Allo Stem Cell Transplantation; Cooking; Physical activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- cooking Education and adapted physical activity (Experimental)
  Interventions: Other: Cooking Education; Other: adapted physical activity

INTERVENTIONS:
Other: Cooking Education — cooking Education and adapted physical activity on patients after allo stem cell transplantation
Other: adapted physical activity — cooking Education and adapted physical activity on patients after allo stem cell transplantation

SUMMARY:
Majority of patients after allo stem cell transplantation have malnutrition and decrease of physical activities. This state impacts on quality of life and on outcome of some complications like infections, graft versus host disease and could decrease the overall survival. In this study, the investigators propose cooking education and adapted physical activity to improve that. Cooking education and adapted physical activity at home will be performed by two famous chefs for the first one and by a sportive coach for the second every twice week.

DETAILED DESCRIPTION:
Bone marrow transplantation is the main strategy to cure leukemia and others hematopoietic malignancies. It includes a first step of chemotherapy during several days (combined sometimes to radiotherapy), a second step of stem cells infusion and a third step of management of complications during several months: side effects, infections or graft versus host disease (GvHD). Symptoms are cutaneous, hepatic and digestive (nausea, diarrhea, vomiting) and could be unfortunately followed by the death of the patients.

Nutritional status is known to be important during the treatment of all cancers. After bone marrow transplantation, patients could have some digestive disorders that could induce malnutrition that could have an impact of time of hospitalization, intensity of complications and outcome of these ones.

When patients go back home after allo stem cell transplantation, they take several medicines, they have digestive side effects of past treatments could alter mucous, taste and all digestive tracts. During at least 100 days, patients take immunosuppressive therapies and they are going to develop new immune system. Therefore, they must follow some food rules to avoid infectious diseases. Patients feel some difficulties to eat good food and refuse often social activities. All of these have an impact on quality of life and induce an increase of malnutrition observed already directly after allo stem cell transplantation. Some complications could also increase malnutrition like digestive GvHD or digestive infections. Malnutrition could also induce physical troubles. Patients need until one year to recover physical conditions before the disease.

The aims of the study are to improve nutritional status and physical activity of patients after allo stem cell transplantation.

The investigators propose at all patients included in the study cooking education and adapted physical activity every twice week in alternance. Cooking education will be performed by two famous chefs in their kitchens. Patients (until 3 months after bone marrow transplantation) and one member of their family are invited to cook and taste. They will receive lot of advice to make several recipes at home and will adapt their cooking methods to respect food rules. Adapted physical activity will be performed by a sportive coach at home. The coach will give them some physical exercises to do between two sessions.

Patients, aged more than 18 years old and signing the consent form, are included in the study before allo stem cell transplantation. Nutritional status evaluation will be performed by a nutritionist using some tests: sit up test, hand grip, bioelectrical impedance analysis, mid upper arm circumference, analogic evaluation of appetite, blood tests: C reactive protein, transthyretin, albumin. The nutritionist will analyze also body mass index, the weight loss percent, the subjective global assessment, the health quality of life assessment.

Evaluation will be performed before allo stem cell transplantation, at day 0, 30, 100 and 300.

The aims of the study are to observe an improvement of nutritional status, quality of life, a decrease of the number of infections and GvHD and at the end an increase of overall survival.

ELIGIBILITY:
Inclusion Criteria:

* Patient at least 18 years old
* Having been an allograft of CSH
* Patient having read and understood the information note related to the study, and signed the informed consent form.

Exclusion Criteria:

* Patient requiring nutritional support by enteral or parenteral route at J30
* Follow-up of the patient considered difficult by the investigator.
* Patient with a linguistic or psychic disability to understand the information.
* Vulnerable patient under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-03-21 (Actual); Primary Completion 2022-05-09 (Actual); Study Completion 2023-02-12 (Actual)

PRIMARY OUTCOMES:
Body mass index | at pre transplant
  Body mass index
Body mass index | at Day 0
  Body mass index
Body mass index | at Day 30
  Body mass index
Body mass index | at Day 100
  Body mass index
Body mass index | at Day 300
  Body mass index
visual analogic scale of appetite | at pre transplant
  It allows a visual assessment, by the patient himself, of his food intake, using an analog scale, or a choice of portions consumed.Visual analog scales (VAS) are reliable tools to evaluate hunger and satiety at point of food consumption. Score from 1 to 10. There are not better or worse values.
visual analogic scale of appetite | at Day 0
  It allows a visual assessment, by the patient himself, of his food intake, using an analog scale, or a choice of portions consumed.Visual analog scales (VAS) are reliable tools to evaluate hunger and satiety at point of food consumption. Score from 1 to 10. There are not better or worse values
visual analogic scale of appetite | at Day 30
  It allows a visual assessment, by the patient himself, of his food intake, using an analog scale, or a choice of portions consumed.Visual analog scales (VAS) are reliable tools to evaluate hunger and satiety at point of food consumption. Score from 1 to 10. There are not better or worse values
visual analogic scale of appetite | at Day 100
  It allows a visual assessment, by the patient himself, of his food intake, using an analog scale, or a choice of portions consumed.Visual analog scales (VAS) are reliable tools to evaluate hunger and satiety at point of food consumption. Score from 1 to 10. There are not better or worse values
visual analogic scale of appetite | at Day 300
  It allows a visual assessment, by the patient himself, of his food intake, using an analog scale, or a choice of portions consumed.Visual analog scales (VAS) are reliable tools to evaluate hunger and satiety at point of food consumption. Score from 1 to 10. There are not better or worse values
sit up test | at pre transplant
  sit up test
sit up test | at Day 0
  sit up test
sit up test | at Day 30
  sit up test
sit up test | at Day 100
  sit up test
sit up test | at Day 300
  sit up test
bio electrical impedance analysis, | at pre transplant
  it's measuring the resistance of biological tissues
bio electrical impedance analysis, | at Day 0
  it's measuring the resistance of biological tissues
bio electrical impedance analysis, | at Day 30
  it's measuring the resistance of biological tissues
bio electrical impedance analysis, | at Day 100
  it's measuring the resistance of biological tissues
bio electrical impedance analysis, | at Day 300
  it's measuring the resistance of biological tissues
hand grip | at pre transplant
  hand grip
hand grip | at Day 0
  hand grip
hand grip | at Day 30
  hand grip
hand grip | at Day 100
  hand grip
hand grip | at Day 300
  hand grip

SECONDARY OUTCOMES:
Quality of life assessment, | at pre transplant
  it's a satisfaction patient's scale
Quality of life assessment, | at Day 0
  it's a satisfaction patient's scale
Quality of life assessment, | at Day 30
  it's a satisfaction patient's scale
Quality of life assessment, | at Day 100
  it's a satisfaction patient's scale
Quality of life assessment, | at Day 300
  it's a satisfaction patient's scale
number of infections, | at pre transplant
  number of infections,
number of infections, | at Day 0
  number of infections,
number of infections, | at Day 30
  number of infections,
number of infections, | at Day 100
  number of infections,
number of infections, | at Day 300
  number of infections,
number of graft versus host disease, | at pre transplant
  number of graft versus host disease,
number of graft versus host disease, | at Day 0
  number of graft versus host disease,
number of graft versus host disease, | at Day 30
  number of graft versus host disease,
number of graft versus host disease, | at Day 100
  number of graft versus host disease,
number of graft versus host disease, | at Day 300
  number of graft versus host disease,
overall survival | at pre transplant
  overall survival
overall survival | at Day 0
  overall survival
overall survival | at Day 30
  overall survival
overall survival | at Day 100
  overall survival
overall survival | at Day 300
  overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Thomas CLUZEAU, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- CHU de Nice - Hôpital de l'Archet, Nice, France